CLINICAL TRIAL: NCT00301821
Title: A Phase II Study of Epratuzumab, Rituximab (ER)-CHOP for Patients With Previously Untreated Diffuse Large B-Cell Lymphoma
Brief Title: Monoclonal Antibody Therapy and Combination Chemotherapy in Treating Patients With Stage II, Stage III, or Stage IV Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0489; NCI-2012-02685 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000459932 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2015-03-24 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — epratuzumab; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epratuzumab + Rituximab + CHOP (Experimental): One arm open label.
  Interventions: Biological: epratuzumab; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: epratuzumab
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Monoclonal antibodies, such as epratuzumab and rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving monoclonal antibody therapy together with chemotherapy may kill more cancer cells.> PURPOSE: This phase II trial is studying how well giving monoclonal antibody therapy together with combination chemotherapy works in treating patients with stage II, stage III, or stage IV diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:> Primary>

* Assess the efficacy of epratuzumab and rituximab in combination with cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone (CHOP), as measured by 12-month, event-free survival, in patients with previously untreated stage II, III, or IV diffuse large B-cell lymphoma.>
* Assess the use of positron emission tomography (PET) scan routinely early in treatment and after completion of treatment.>
* Assess the functional response rate (complete response, partial response, or stable disease by CT scan and PET negative) in patients treated with this regimen.>
* Assess the safety of this treatment regimen.> Secondary>
* Correlate laboratory prognostic factors for large cell lymphoma with clinical response to this regimen.> OUTLINE: This is a multicenter study.> Patients receive epratuzumab IV over 1 hour on day 1, rituximab IV over 4-8 hours on day 1 or days 1 and 2, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1 or 2, and oral prednisone on days 1-5 or 2-6. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.> After completion of study treatment, patients are followed periodically for up to 5 years.> PROJECTED ACCRUAL: A total of 86 patients will be accrued for this study.>

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell lymphoma

  * B-cell phenotype (CD20+) as determined by immunohistochemistry (IHC) or flow cytometry
  * Stage II, III, or IV disease
* CD22+ tumor by IHC*

NOTE: *CD22 status may be determined after study enrollment

* Measurable disease, defined as at least 1 lesion ≥ 1.5 cm by CT scan or physical exam
* No relapsed or refractory non-Hodgkin's lymphoma
* No history of transformed lymphoma
* No CNS lymphoma

  * CNS symptoms or bone marrow or sinus involvement must have absence of CNS lymphoma confirmed by lumbar puncture

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-3

  - For patients with ECOG PS 3, the PS must be disease related
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 2 mg/dL (if total bilirubin > 2 mg/dL, direct bilirubin should be within normal limits)
* AST ≤ 3 times upper limit of normal (ULN) (5 times ULN if there is liver involvement)
* Creatinine ≤ 2 times ULN
* Life expectancy ≥ 12 weeks
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* No active serious infection requiring antibiotics
* No New York Heart Association class III or IV heart disease
* No other primary malignancy within the past 5 years, except for squamous cell or basal cell carcinoma of the skin, in situ carcinoma of the cervix, or previously treated prostate cancer with a stable prostate-specific antigen
* No known HIV positivity
* No known hepatitis B or C infection
* Ejection fraction ≥ 45% by MUGA or echocardiogram (required if patients has a history of heart disease or is ≥ 50 years old)
* Willing to provide blood and tissue samples for mandatory translational research component of study

PRIOR CONCURRENT THERAPY:

* No prior therapy for diffuse large B-cell lymphoma, including the following:

  * Chemotherapy
  * Immunotherapy
  * Biologic therapy
  * Radiotherapy
* Prior short course (≤ 14 days) of corticosteroids allowed
* Prior splenectomy allowed
* No prior pelvic irradiation
* No other concurrent investigational agents
* No concurrent chemotherapy, immunotherapy, or radiotherapy
* No concurrent enrollment on another treatment study involving a pharmacologic agent (e.g., drugs, biologics, immunotherapy, or gene therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Micallef, MD, Study Chair — Mayo Clinic
Locations (162):
- United States (162):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital and Medical Center, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Hematology-Oncology Associates of Fredericksburg, Incorporated, Fredericksburg, Virginia
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin

REFERENCES:
- [Background] Micallef IN, Kahl BS, Maurer MJ, Dogan A, Ansell SM, Colgan JP, Geyer S, Inwards DJ, White WL, Habermann TM. A pilot study of epratuzumab and rituximab in combination with cyclophosphamide, doxorubicin, vincristine, and prednisone chemotherapy in patients with previously untreated, diffuse large B-cell lymphoma. Cancer. 2006 Dec 15;107(12):2826-32. doi: 10.1002/cncr.22342. PMID 17099879
- [Result] Maurer MJ, Micallef IN, Cerhan JR, Katzmann JA, Link BK, Colgan JP, Habermann TM, Inwards DJ, Markovic SN, Ansell SM, Porrata LF, Johnston PB, Nowakowski GS, Thompson CA, Gupta M, Syrbu SI, Kurtin PJ, Macon WR, Nikcevich DA, Witzig TE. Elevated serum free light chains are associated with event-free and overall survival in two independent cohorts of patients with diffuse large B-cell lymphoma. J Clin Oncol. 2011 Apr 20;29(12):1620-6. doi: 10.1200/JCO.2010.29.4413. Epub 2011 Mar 7. PMID 21383282
- [Result] Micallef IN, Maurer MJ, Wiseman GA, Nikcevich DA, Kurtin PJ, Cannon MW, Perez DG, Soori GS, Link BK, Habermann TM, Witzig TE. Epratuzumab with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone chemotherapy in patients with previously untreated diffuse large B-cell lymphoma. Blood. 2011 Oct 13;118(15):4053-61. doi: 10.1182/blood-2011-02-336990. Epub 2011 Jun 14. PMID 21673350
- [Result] Micallef IN, Maurer MJ, Nikcevich DA, et al.: Final results of NCCTG N0489: epratuzumab and rituximab in combination with cyclophosphamide, doxorubicin, vincristine, and prednisone chemotherapy (ER-CHOP) in patients with previously untreated diffuse large B-cell lymphoma. [Abstract] J Clin Oncol 27 (Suppl 15): A-8508, 2009.
- [Derived] Ghesquieres H, Larrabee BR, Haioun C, Link BK, Verney A, Slager SL, Ketterer N, Ansell SM, Delarue R, Maurer MJ, Fitoussi O, Habermann TM, Peyrade F, Dogan A, Molina TJ, Novak AJ, Tilly H, Cerhan JR, Salles G. FCGR3A/2A polymorphisms and diffuse large B-cell lymphoma outcome treated with immunochemotherapy: a meta-analysis on 1134 patients from two prospective cohorts. Hematol Oncol. 2017 Dec;35(4):447-455. doi: 10.1002/hon.2305. Epub 2016 Jun 10. PMID 27282998
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this study 107 patients with newly diagnosed diffuse large B-cell lymphoma (DLBCL) were enrolled. Twenty-six (24%) patients were declared ineligible based on pathology review; 1 patient canceled before beginning treatment.
Groups:
- Epratuzumab + Rituximab + CHOP: One arm open label. Epratuzumab, Rituximab, Cyclophosphamide, Doxorubicin hydrochloride, Prednisone, Vincristine sulfate
Period: Overall Study
Arm/Group | Epratuzumab + Rituximab + CHOP
Started | 107
Completed | 81
Not Completed | 26
Not completed — Ineligible | 25
Not completed — Cancel | 1

BASELINE CHARACTERISTICS:
Groups:
- Epratuzumab + Rituximab + CHOP: One arm, open label. Epratuzumab, Rituximab, Cyclophosphamide, Doxorubicin hydrochloride, Prednisone, Vincristine sulfate.
Arm/Group | Epratuzumab + Rituximab + CHOP
Number analyzed (Participants) | 107
Age, Continuous [Median (Full Range); unit: years] | 62 [21 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 59
Region of Enrollment [Number; unit: participants]
  United States | 107

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival After 12 Months
Description: The primary endpoint of the trial was the percentage of the eligible patients who were alive and event-free 12 months after enrollment to the study (EFS12).
Time Frame: From Baseline to 12 months
Population: First 76 eligible participants were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Epratuzumab + Rituximab + CHOP
Number analyzed (Participants) | 76
percentage of participants | 78

2. Secondary Outcome: Overall Survival
Description: Percentage of participants alive at different time points
Time Frame: time from study entry to 36 months
Population: Intent To Treat (All Patients)
Measure: Number; unit: percentage of Participants
Arm/Group | Epratuzumab + Rituximab + CHOP
Number analyzed (Participants) | 107
percentage of Participants
  Overall Survival at 12 months | 89
  Overall Survival at 24 months | 81
  Overall Survival at 36 months | 80

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Percentage of participants Progression-free at different time points. Response was assessed using International Workshop Response Criteria.38 Response is based on CT alone. Relapse or progression is defined as Enlarging liver/spleen, new sites, New or increased lymph nodes, New or Increased lymph node masses, bone marrow reappearance.
Time Frame: the time from study entry to 36 months
Population: Intent To Treat (All Patients)
Measure: Number; unit: percentage of participants
Arm/Group | Epratuzumab + Rituximab + CHOP
Number analyzed (Participants) | 107
percentage of participants
  Progression Free Survival at 12 months | 85
  Progression Free Survival at 24 months | 77
  Progression Free Survival at 36 months | 76

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate will be estimated by the number of patients with objective status of partial response (PR), unconfirmed complete response (CRu), or complete response (CR) during the first 6 cycles of treatment divided by number of evaluable patients (met eligibility criteria, signed consent form, and started treatment). Response was assessed using International Workshop Response Criteria.38 Response is based on CT alone. Relapse or progression is defined as Enlarging liver/spleen, new sites, New or increased lymph nodes, New or Increased lymph node masses, bone marrow reappearance.
Time Frame: Baseline to first 6 cycles of treatment
Population: Out of the 107 patients enrolled, Twenty-five patients were declared ineligible based on pathology review; 1 patient canceled before beginning treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Epratuzumab + Rituximab + CHOP
Number analyzed (Participants) | 81
percentage of participants | 95

ADVERSE EVENTS:
Description: One patient canceled before beginning treatment.
Arm/Group | Epratuzumab + Rituximab + CHOP
Serious Adverse Events (participants affected / at risk) | 72/106
Other Adverse Events (participants affected / at risk) | 105/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epratuzumab + Rituximab + CHOP (N=106)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (16)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (8)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Cecal hemorrhage (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Gastic fistula (Gastrointestinal disorders) | 1 (1)
Ileal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Leukocyte count decreased (Investigations) | 62 (136)
Lymphocyte count decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 67 (149)
Platelet count decreased (Investigations) | 9 (10)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epratuzumab + Rituximab + CHOP (N=106)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (9)
Hemoglobin decreased (Blood and lymphatic system disorders) | 30 (68)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 9 (12)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (6)
Ileus (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 9 (11)
Nausea (Gastrointestinal disorders) | 12 (17)
Oral pain (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 28 (47)
Chest pain (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 36 (89)
Fever (General disorders) | 2 (2)
General symptom (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 14 (14)
Hypersensitivity (Immune system disorders) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 2 (2)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Gastric infection (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 3 (4)
Infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Skin infection (Infections and infestations) | 3 (3)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral hepatitis (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Leukocyte count decreased (Investigations) | 88 (326)
Lymphocyte count decreased (Investigations) | 7 (23)
Neutrophil count decreased (Investigations) | 78 (200)
Platelet count decreased (Investigations) | 71 (260)
Weight gain (Investigations) | 3 (10)
Weight loss (Investigations) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 9 (12)
Blood glucose increased (Metabolism and nutrition disorders) | 18 (32)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (6)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (8)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (8)
Headache (Nervous system disorders) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (2)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 50 (199)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 4 (4)
Bladder obstruction (Renal and urinary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (2)
Kidney pain (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 40 (150)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Sweating (Skin and subcutaneous tissue disorders) | 2 (4)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Thrombosis (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes